CLINICAL TRIAL: NCT01731587
Title: Phase Ib, Single-arm, Proof-of-principle Trial Investigating the Cytokine Profile and Specific T Cell Response in Peripheral Blood of Non-small Cell Lung Cancer (NSCLC) Subjects With Unresected Stage III Disease Treated With L-BLP25
Brief Title: Anti-cancer MUC1-specific Immunotherapy for Unresectable Stage III Non-small Cell Lung Cancer
Acronym: FINGERPRINT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The objectives of this trial are no longer deemed appropriate for the clinical development of L-BLP25 therefore this trial is withdrawn
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EMR 63325-019; 2012-001435-31 (EudraCT Number)
Record Dates: First submitted 2012-10-11; First posted 2012-11-22 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC) Stage III
Keywords: Non-small cell lung cancer (NSCLC); exploratory study; L-BLP25
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-BLP25 plus Cyclophosphamide (CPA) (Experimental)
  Interventions: Other: Biological: MUC1 peptide specific immunotherapy; Drug: Cyclophosphamide (CPA)

INTERVENTIONS:
Other: Biological: MUC1 peptide specific immunotherapy — Eight consecutive weekly subcutaneous administration with reconstituted L-BLP25 (containing 806 microgram of BLP25 lipopeptide) followed by administrations at 6-week intervals, commencing at Week 14, until disease progression is documented.
  Other Names: EMD531444; Stimuvax®
Drug: Cyclophosphamide (CPA) — A single intravenous infusion of 300 milligram per square meter (to a maximum of 600 milligram) of CPA will be given three days before the first L-BLP25 administration.
  Other Names: L01AA01; Endoxana

SUMMARY:
Phase Ib study investigating whether liposome BLP25 mucin-1 (MUC1) peptide-specific immunotherapy (L-BLP25) administered as weekly subcutaneous doses over 8 weeks following a single dose of intravenous cyclophosphamide (CPA) induces a reproducible cytokine pattern measured in the serum of unresected Stage III non-small cell lung cancer (NSCLC) subjects after first-line chemo-radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented unresectable Stage III NSCLC, as defined by American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC) 7th edition (2009) criteria. All histological subtypes are acceptable, including bronchioalveolar carcinomas
* Documented stable disease or objective response, according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.0, after primary chemo-radiotherapy (either sequential or concomitant) for unresected Stage III disease, within 4 weeks (28 days) prior to enrollment
* Receipt of concomitant or sequential chemo-radiotherapy, consisting of a minimum of two cycles of platinum-based chemotherapy and a minimum radiation dose of greater than equal to 50 Gray. Subjects must have completed the primary thoracic chemo-radiotherapy at least 4 weeks (28 days) and no later than 84 days prior to enrollment. Subjects who received prophylactic brain irradiation as part of primary chemo-radiotherapy are eligible
* Platelet count greater than or equal to 140 * 10^9 per liter, white blood cell (WBC) greater than or equal to 2.5 * 10^9 per liter, and hemoglobin greater than or equal to 90 gram per liter
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1

Additional Inclusion Criteria apply

Exclusion Criteria:

* Pre-therapies:

  * Previous lung cancer specific therapy (including surgery) other than primary chemo-radiotherapy
  * Receipt of immunotherapy within 4 weeks (28 days) prior to enrollment. Note: Subjects who have received monoclonal antibodies for imaging are acceptable
  * Receipt of investigational systemic drugs (including off-label use of approved products) within 4 weeks (28 days) prior to enrollment
* Disease status:

  * Metastatic disease
  * Malignant pleural effusion at initial diagnosis and/or at trial entry
  * Past or current history of neoplasm other than lung carcinoma, except for curatively treated nonmelanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
  * Autoimmune disease
  * A recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary or congenital immunodeficiencies
  * Any preexisting medical condition requiring systemic chronic steroid or immunosuppressive therapy (steroids for the treatment of radiation pneumonitis are allowed)
  * Known Hepatitis B and/or C
  * Active infection at enrollment, including but not limited to, flu-like infections, urinary tract infections, bronchopulmonary infections, etc
* Physiological functions:

  * Clinically significant hepatic dysfunction (that is, alanine aminotransferase [ALT] greater than 2.5 times normal upper limit [ULN]; or aspartate aminotransferase [AST] greater than 2.5 times ULN; or bilirubin greater than or equal to 1.5 * ULN)
  * Clinically significant renal dysfunction (that is, serum creatinine greater than or equal to 1.5 * ULN)
  * Clinically significant cardiac disease, for example, New York Heart Association (NYHA) Classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months as confirmed by an electrocardiogram (ECG)
  * Splenectomy
  * Infectious process that in the opinion of the investigator could compromise the subject's ability to mount an immune response

Additional Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-01

PRIMARY OUTCOMES:
Immune response defined as change from baseline in serum cytokine levels after L-BLP25 administration at Week 1, 4 and 8 | Pre-dose (Day -3) up to 24 hours after L-BLP25 administration at Week 1, 4 and 8

SECONDARY OUTCOMES:
Evaluation of a cellular immune response following treatment with L-BLP25 | Pre-dose (Day -3) and at 24 hours after L-BLP25 administration at Week 4 and 8
Change from baseline in alternative immune or inflammatory serum soluble immune mediators such as interferon alpha (IFNα), transforming growth factor beta (TGFβ), or C-reactive protein (CRP) at 6, 12, and 24 hours after L-BLP25 administration. | Pre-dose (Day -3) up to 24 hours after L-BLP25 administration at Week 1, 4 and 8
Number of subjects with adverse events (AEs) | Up to 6 weeks after the last dose of L-BLP25

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck KGaA, Darmstadt, Germany

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562